CLINICAL TRIAL: NCT02779088
Title: Department of Physical Medicine and Rehabilitation,National Taiwan University Hosptial,Bei-Hu Brance and National Taiwan University College of Medicine,Taipei,Taiwan
Brief Title: The Physical Fitness Cohort Study in the Community-dwelling Elderly in the WanHwa Area.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201601091RIND
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia
Keywords: physical fitness,body composition,sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Exercise; Nutritional Status

STUDY DESIGN:
Intervention Model Description: The investigators invited around 60 persons with sarcopenia by telephone to attend the study and randomly assigned them to group A and B (around 30 persons in each). Group A first accepted exercise and nutrition intervention and then was given the education course. Group B was treated in the reversed order.
Masking Description: Participants and investigator don't know which group the participants are assigned to before randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early exercise and nutrition (Experimental): Enrolled participants with sarcopenia will be randomized to receive either strengthening exercise and nutrition or education courses (DVD and handbook) first and then will receive the opposite intervention subsequently. The study will consist of two periods of 12 weeks separated by a washout period of 2 weeks. It's the AB/BA study. Subjects in the AB arm receive exercise and nutrition intervention first, followed by the education course.
  Interventions: Other: exercise and nutrition
- Delayed exercise and nutrition (Active Comparator): Enrolled participants with sarcopenia will be randomized to receive either strengthening exercise and nutrition or education courses (DVD and handbook) first and then will receive the opposite intervention subsequently. The study will consist of two periods of 12 weeks separated by a washout period of 2 weeks. It's the AB/BA study. Subjects in the BA arm receive the education course first, followed by exercise and nutrition.
  Interventions: Other: exercise and nutrition

INTERVENTIONS:
Other: exercise and nutrition — Exercise:muscle strengthening exercise Nutrition: 7.2 g branched chain amino acid every day and 1200 mg Ca+800 IU Vitamin D3

SUMMARY:
The aims of this study are to establish the cohort of elder population based on parameters of health-related fitness, body compositions, blood biochemistry, blood biomarker, balance, quality of life, and musculoskeletal ultrasonography; and to evaluate the association between fitness parameters and disease incidence with those data.

DETAILED DESCRIPTION:
The aims of this study are to establish the cohort of elder population based on parameters of health-related fitness, body compositions, blood biochemistry, blood biomarker, balance, quality of life, and musculoskeletal ultrasonography and to evaluate the association between fitness parameters and disease incidence with these data. We expect to recruit 1200 adults who attend the annual health check-up in National Taiwan University, BeiHu Branch in 2016 and 2017 and to train 60 individuals having sarcopenia with strengthening exercise. This study will establish the urban elderly cohort, measure both physical and functional parameters, find the risk factors for aging, and validate the role of strength training for those sarcopenia patients. We hope this study will be widely cited in related fields in the future.

ELIGIBILITY:
Inclusion criteria:

The investigators are ready to find out the individuals aged above 65 years and having sarcopenia. The 60 individuals must be evaluated their physical fitness in advance. The investigators plan to perform exercise and nutrition intervention for the individuals.

Exclusion criteria:

1. Patients with heart rhythm, atrial fibrillation, ventricular bigeminy, infections, tumors, and blood disease,etc.
2. Individuals has lived in nursing home or long-term care institutions.
3. Individuals cannot stand steadily. 4 Individuals cannot fill the questionnaires by his own.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-04-24 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Change from skeletal muscle mass,grip and pace between the baseline, 1st follow-up (12 weeks) and 2nd follow-up (26 weeks) after the whole intervention process | At the baseline, 1st follow-up (12 weeks) and 2nd follow-up (26 weeks) after the whole intervention process
  Skeletal muscle mass,grip and pace were assessed the baseline, 1st follow-up (12 weeks) and 2nd follow-up (26 weeks) after the whole intervention process

SECONDARY OUTCOMES:
Change from telomere's length at the baseline, 1st follow-up (12 weeks) and 2nd follow-up (26 weeks) after the whole intervention process | At the baseline, either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process
  The investigators want to measure the change of telomere's length at the baseline and , either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process
Change of Terra RNA, physical fitness and other components of body compositions at the baseline, either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process | at the baseline, either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process
  The investigators want to measure the correlation of Terra RNA with physical fitness and other components of body compositions.
the difference of ECV at the baseline, 1st follow-up (12 weeks) and 2nd follow-up (26 weeks) after the whole intervention process | At the baseline, either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process
  The investigators want to measure the difference of ECV at the baseline, either at 1st follow-up (12 weeks) or 2nd follow-up (26 weeks) after the whole intervention process

CONTACTS AND LOCATIONS:
Overall Officials: Der-Sheng Han MD, PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital BeiHu Brance,Taipei
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang KV, Wu WT, Huang KC, Han DS. Effectiveness of early versus delayed exercise and nutritional intervention on segmental body composition of sarcopenic elders - A randomized controlled trial. Clin Nutr. 2021 Mar;40(3):1052-1059. doi: 10.1016/j.clnu.2020.06.037. Epub 2020 Jul 14. PMID 32723507